CLINICAL TRIAL: NCT00074191
Title: Combination Chemotherapy (Methotrexate, Procarbazine And CCNU), Intraventricular Cytarabine And Methotrexate, +/- Intra-Ocular Chemotherapy For Patients With Primary Central Nervous System Lymphoma
Brief Title: Methotrexate, Procarbazine, Lomustine, Dexamethasone, and Cytarabine in Treating Patients With Primary CNS Lymphoma
Acronym: Protocol-A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Masking: None | Purpose: Treatment
Other Study IDs: IRB00000929; 5729-1 (Other: OHSU IRB (discontinued number)); ONC-99054-1 (Other: OHSU Knight Cancer Institute); 929 (Other: OHSU eIRB); OHSU-5729-1 (Other: OHSU IRB (legacy number))
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Lymphoma
Keywords: intraocular lymphoma; primary central nervous system lymphoma
MeSH Terms: conditions — Lymphoma; Intraocular Lymphoma | interventions — Cytarabine; Dexamethasone; Lomustine; Methotrexate; Procarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cytarabine
Drug: dexamethasone
Drug: lomustine
Drug: methotrexate
Drug: procarbazine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as methotrexate, procarbazine, lomustine, dexamethasone, and cytarabine, use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have primary CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity and efficacy of methotrexate, procarbazine, lomustine, dexamethasone, and cytarabine in patients with primary CNS lymphoma.

Secondary

* Determine the ability to recruit adequate numbers of patients for this study.
* Compare progression-free and dementia-free survival with standard measures of overall survival, progression-free survival, disease-free survival, complete response rate, cognitive function, and quality of life of patients treated with this regimen.
* Determine the feasibility of conducting a future phase III study of this treatment regimen in these patients.
* Correlate neuropsychological outcomes with neuroimaging (MRI) outcomes in patients treated with this regimen.

OUTLINE: This is a nonrandomized, multicenter study.

* Induction chemotherapy: Patients receive methotrexate IV over 3 hours on days 1, 10, and 20 and intraventricularly or intrathecally (IT) over 5 minutes on days 1, 5, 10, and 15; oral procarbazine on days 1-7; oral lomustine on day 1; oral dexamethasone every 6 hours on days 1-14 followed by a taper (as tolerated); and cytarabine intraventricularly or IT over 5 minutes on days 1, 5, 10, and 15. Treatment repeats every 42 days for a total of 3 courses. Patients with intraocular lymphoma also receive methotrexate intravitreally twice weekly until the vitreous is clear of cells by slit lamp exam. Patients with stable or responding disease proceed to maintenance therapy.
* Maintenance chemotherapy: Patients receive methotrexate IV over 3 hours and IT over 5 minutes on day 1; oral procarbazine on days 1-7; oral lomustine on day 1; oral dexamethasone every 6 hours on days 1-14 followed by a taper (as tolerated); and cytarabine intraventricularly or IT over 5 minutes on day 1. Treatment repeats every 42 days for a total of 5 courses.

Patients with intraocular lymphoma also receive methotrexate intravitreally weekly for 1 month and then monthly for 1 year.

Quality of life is assessed at baseline, at 6 months, at the completion of treatment, every 6 months for 2 years, and then annually thereafter.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 180 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed intermediate- or high-grade primary CNS lymphoma documented by brain biopsy or cerebrospinal fluid or vitrectomy analysis
* Diagnosed within the past 90 days
* No systemic lymphoma NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 16 to 75

Performance status

* ECOG 0-3 OR
* Karnofsky 40-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 2,500/mm^3
* Hematocrit at least 25% (transfusion allowed)
* Absolute granulocyte count at least 1,200/mm^3
* Platelet count at least 100,000/mm^3 OR at least lower limit of normal (transfusion independent)

Hepatic

* Bilirubin no greater than 2.0 times upper limit of normal

Renal

* Creatinine clearance at least 30 mL/min

Cardiovascular

* Adequate cardiac function to tolerate general anesthesia

Pulmonary

* Adequate pulmonary function to tolerate general anesthesia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 2 months before and during study participation
* No other uncontrolled, clinically significant confounding medical condition within the past 30 days
* No known allergy to study agents
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)

  * Single-agent methotrexate administered within the past 14 days allowed

Endocrine therapy

* Not specified

Radiotherapy

* No prior cranial or spinal radiotherapy

Surgery

* Prior surgery or biopsy allowed

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2000-01; Primary Completion 2000-10 (Actual); Study Completion 2000-10 (Actual)

PRIMARY OUTCOMES:
Survival as measured by clinical and radiographic response at 5 years following completion of study treatment | 5 years

SECONDARY OUTCOMES:
Overall survival as measured by clinical and radiographic response | 5 years
Progression-free survival as measured by clinical and radiographic response until tumor progression | 5 years
Quality of Life (QOL) as measured by EORTC QOL before and after study treatment, every 6 months for 2 years, and then annually | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward A. Neuwelt, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Oregon Health & Science University Cancer Institute, Portland, Oregon, United States